CLINICAL TRIAL: NCT07138339
Title: Radicle Menstrual Wellness™ CSP: A Randomized, Double-Blind, Placebo-Controlled, Trial Evaluating Plant-Based Health and Wellness Products on Menstrual Wellness in Premenopausal Women
Brief Title: Radicle Menstrual Wellness™ CSP: A Trial Evaluating Plant-Based Health and Wellness Products on Menstrual Wellness in Premenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX_C_2506_SP
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Menstrual Wellness

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on their age, menstrual pain, and health outcome score during enrollment then randomized to one of the study arms. Each participant will have an equal chance of being assigned to each study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator): Menstrual Wellness Product Control
  Interventions: Dietary Supplement: Menstrual Wellness Product Placebo Control
- Active Product 1 (Experimental): Menstrual Wellness Product 1
  Interventions: Dietary Supplement: Menstrual Wellness Product 1

INTERVENTIONS:
Dietary Supplement: Menstrual Wellness Product Placebo Control — Participants will use their Menstrual Wellness Product Placebo Control as directed for a period of 12 weeks
  Arms: Placebo Control
Dietary Supplement: Menstrual Wellness Product 1 — Participants will use their Menstrual Wellness Product 1 as directed for a period of 12 weeks
  Arms: Active Product 1

SUMMARY:
A randomized, double-blind, placebo-controlled, trial evaluating plant-based health and wellness products on menstrual wellness in premenopausal women

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants (1) are female, (2) are premenopausal, (3) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome, and (4) express acceptance in taking study products and not knowing the formulation identities until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and women who are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 13 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, at least 21 years old at the time of electronic consent, inclusive of all ethnicities, races, and gender identities
* Assigned sex at birth is female
* Resides in the United States
* Identifies menstrual status as premenopausal
* Reports an average menstrual cycle length of 3 - 6 weeks
* Has the opportunity for at least 30% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.

  -- NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.

  -- Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products and/or pose a safety risk to participants
* Reports an allergy to and/or disinterest in any of the possible study product ingredients
* Lack of reliable daily access to the internet

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Change in Menstrual Distress | 13 weeks
  Difference between rates of change over time in Menstrual Distress as assessed by MEDI-Q (scale 0-125; higher scores = worse menstrual distress)

SECONDARY OUTCOMES:
Change in Wellbeing | 13 weeks
  Difference between rates of change over time in Wellbeing as assessed by WHO-5 (scale 0-25; higher scores = better wellbeing)
Change in Pain Interference | 13 weeks
  Difference in rates of change over time in pain interference score as assessed by PROMIS Pain Interference 6A (scale 6-30; with higher scores corresponding to more severe pain interference)
Change in Pain Intensity | 13 weeks
  Difference in rates of change over time in pain intensity score as assessed by PROMIS Pain Intensity 3A (scale 3-15; with higher scores corresponding to more severe pain intensity)

OTHER OUTCOMES:
Minimal clinical importance difference (MCID) in Menstrual Wellness | 13 weeks
  Likelihood of achieving an MCID in menstrual wellness, as measured by MEDI-Q (scale 0-125; higher scores = worse menstrual wellbeing)
Minimal clinically important difference (MCID) in pain intensity | 13 weeks
  Likelihood of experiencing minimal clinically important difference in pain intensity, as assessed by PROMIS Pain Intensity 3A (scale 3-15; with higher scores corresponding to more severe pain intensity)
Minimal clinical importance difference (MCID) in Wellbeing | 13 weeks
  Likelihood of achieving an MCID in Wellbeing, as measured by WHO-5 (scale 0-25; higher scores = better wellbeing)
Minimal clinically important difference (MCID) in pain interference | 13 weeks
  Likelihood of experiencing minimal clinically important difference in pain interference, as measured by PROMIS Pain interference (6-30; where lower scores indicate less pain interference).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science Inc., Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Related Info — https://www.radiclescience.com